CLINICAL TRIAL: NCT04727151
Title: A Phase 1/2 Trial Investigating the Safety and Efficacy of Autologous TAC T Cell Monotherapy, and TAC T Cells in Combination With Pembrolizumab, in Relapsed HER2-Positive Solid Tumors
Brief Title: TAC T-cells for the Treatment of HER2-positive Solid Tumors
Acronym: TACTIC-2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated by Sponsor for commercial reasons
Sponsor: Triumvira Immunologics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAC01-HER2-03; KEYNOTE-E77 (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: HER2 Positive Gastric Cancer; Metastatic HER2 Positive Gastroesophageal Junction Cancer
Keywords: HER2 Positive Gastric Cancer; HER2 Positive gastroesophageal adenocarcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: In Phase 1, escalating doses of TAC01-HER2 will be evaluated to identify the RP2D of the monotherapy arm and the combination arm using the classic keyboard design. In Phase 2, dose expansion groups will further evaluate the safety, efficacy, and PK of the MTD or RP2D for TAC01-HER2 as a monotherapy and in combination with pembrolizumab in subjects with gastric and gastroesophageal adenocarcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAC01-HER2 (Experimental): Lymphodepletion followed by TAC01-HER2 as a single IV infusion, with a potential for a second dose administration.
  Interventions: Biological: TAC01-HER2
- TAC01-HER2 plus pembrolizumab (Experimental): Lymphodepletion followed by TAC01-HER2 as a single IV infusion, followed by pembrolizumab administration.
  Interventions: Biological: TAC01-HER2 plus pembrolizumab

INTERVENTIONS:
Biological: TAC01-HER2 — TAC01-HER2 and:
  * fludarabine and cyclophosphamide, or
  * clofarabine and cyclophosphamide, or
  * bendamustine, or
  * cyclophosphamide
  Arms: TAC01-HER2
Biological: TAC01-HER2 plus pembrolizumab — TAC01-HER2 plus pembrolizumab and:
  * fludarabine and cyclophosphamide, or
  * clofarabine and cyclophosphamide, or
  * bendamustine, or
  * cyclophosphamide
  Other Names: Keytruda
  Arms: TAC01-HER2 plus pembrolizumab

SUMMARY:
TAC01-HER2 is a novel cell therapy that consists of genetically engineered autologous T cells expressing T-cell Antigen Coupler (TAC) that recognizes human epidermal growth factor receptor 2 (HER2). TAC directs T-cells to the targeted antigen (HER2), and once engaged with the target, activates them via the endogenous T cell receptor.

This is an open-label, multicenter Phase 1/2 study that aims to establish safety, maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D), pharmacokinetic profile and efficacy of TAC01-HER2 as a monotherapy, and in combination with pembrolizumab, in subjects with HER2 positive gastric and gastroesophageal adenocarcinoma.

DETAILED DESCRIPTION:
The TAC technology is a novel approach to modifying T cells, herein referred to as TAC T cells, and using them in the treatment of solid tumors. TAC T cells are produced through genetic engineering, incorporating TAC receptors into a patient's own T cells. This redirects these enhanced T cells to specific cancer antigens, and upon recognition, activates them through the natural signaling pathways of the endogenous TCR. In the TAC01-HER2 engineered T cell product; TAC T cells recognize the HER2 protein present on the surface of tumor cells, and eradicate them. Consequently, it is hypothesized TAC01-HER2 will be potentially safe and effective in treating patients with HER2+ solid tumors and provide a clinically meaningful therapeutic benefit in patient populations with high unmet medical need.

This is a first-in-human study investigating TAC01-HER2 to evaluate the safety, MTD or RP2D, PK, and efficacy in subjects with HER2+ solid tumors who have been treated after at least 2 lines of prior therapy in Phase 1 and after at least 2 lines and no more than 4 lines of prior therapy in Phase 2.

In Phase 1, escalating doses of TAC01-HER2 will be evaluated to identify the RP2D using the classic keyboard design method. The monotherapy arm will treat all subjects with HER2-positive solid tumors that meet the eligibility criteria (completed). The combination arm will treat all 2+ or 3+ HER2-positive subjects with gastric or gastroesophageal AC who meet the eligibility criteria.

In Phase 2, dose expansion groups will further evaluate the efficacy, safety, and PK of the MTD or RP2D for TAC01-CLDN18.2 in subjects with gastric and esophageal adenocarcinoma. In Phase 2, a Simon 3-stage design will be used to enroll up to 36 subjects in Group A (monotherapy arm) and 34 subjects in Group B (combination arm).

In summary:

* Phase I monotherapy arm: Dose escalation in any HER2-positive solid tumor (completed).
* Phase I combination therapy arm: Dose escalation in combination with pembrolizumab in 2+ or 3+ HER2-positive gastric and gastroesophageal adenocarcinoma
* Phase II: Dose expansion cohorts: 2+ or 3+ HER2-positive gastric or gastroesophageal adenocarcinoma treated with TAC01-HER2 as a monotherapy (Group A) or in combination with pembrolizumab (Group B).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age ≥ 18 years at the time of informed consent.
3. For Phase 1 and Phase 2:

   * Phase 1 monotherapy (completed): HER2 1+, 2+, 3+ by IHC by central laboratory confirmation
   * Phase 1 combination therapy and Phase 2: HER2 2+, 3+ by IHC and FISH by central laboratory confirmation
4. Histologically confirmed advanced, metastatic, unresectable solid tumors (regardless of PD-L1 expression levels; Phase 1 monotherapy) and histologically confirmed advanced, metastatic, unresectable gastric or esophageal adenocarcinoma (regardless of PD-L1 expression levels for Phase 1 combination therapy and Phase 2) after at least 2 prior lines of therapy (Phase 1) or after at least 2 and no more than 4 prior lines of therapy (Phase 2).

   1. HER2+ incurable malignancies for which no standard-of-care HER2 targeted therapy exists may be enrolled regardless of the number of prior treatment lines, as long as in the opinion of the investigator the subject would be unlikely to tolerate or derive clinically meaningful benefit from other available treatment options.
   2. For breast cancer subjects, both prior lines of therapy must have included HER2-targeted agents per current standard-of-care.
   3. Subjects with solid tumors with genetic alterations and mutations (such as BRAF, BRCA, EGFR mutations, and ALK translocation) where approved targeted therapies were available to their specific cancers must have been previously treated with such approved therapies or refused such approved targeted therapy for their cancers prior to enrollment, or in the opinion of the investigator would be unlikely to tolerate or derive clinically meaningful benefit from these standard-of-care therapies.
5. Measurable disease per RECIST 1.1 at time of enrollment.
6. ECOG performance status of 0 or 1 at Screening.
7. Life expectancy of at least 12 weeks.
8. Adequate organ and bone marrow reserve function.
9. Recovery to Grade ≤1 or Baseline for any toxicities due to previous therapy.
10. Adequate vascular access for leukapheresis.
11. Negative pregnancy test and use of highly effective contraception.
12. Undetectable HBV viral load.
13. HCV viral load is undetectable.

Exclusion Criteria:

1. Intolerant to any component of TAC01-HER2.
2. Prior treatment with any of the following:

   1. Adoptive cell transfer of any kind, including CAR T cells
   2. Gene therapy
3. Investigational medicinal product within 5 half-lives or 21 days prior to leukapheresis, whichever is shorter.
4. Receipt of a live or live-attenuated vaccine within 30 days prior to study treatment.
5. Monoclonal antibody (mAb), including PD-1 and PD-L1, therapies within 21 days prior to leukapheresis.
6. Radiation within 28 days prior to enrollment. Palliative radiation is allowed up to 14 days prior to enrollment if non-irradiated lesions are present.
7. Chemotherapy or targeted small molecule therapy within 14 days prior to leukapheresis, or within 7 days prior to leukapheresis for erlotinib, gefitinib, afatinib, or crizotinib.
8. Colony stimulating factors, including granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), erythropoietin, and other hematopoietic cytokines, within 14 days prior to leukapheresis.
9. Immunosuppressive medication within 14 days or corticosteroid treatment < 72 hours prior to enrollment.
10. History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. (Brain metastasis - non-progressive or previously treated and currently stable - are permitted.)
11. Active inflammatory neurological disorders (e.g., Guillain-Barre Syndrome, amyotrophic lateral sclerosis, multiple sclerosis).
12. Active autoimmune disease (e.g., lupus, rheumatoid arthritis, Sjogren's syndrome) requiring systemic disease modifying agents in the past 2 years.
13. Active or uncontrolled hepatitis B or C (HCV ribonucleic acid [RNA] positive) infection or any history of or active human immunodeficiency virus (HIV) infection.
14. Uncontrolled, acute, or life-threatening bacterial, viral, or fungal infection. Subjects with ongoing use of prophylactic antibiotics, antifungals, or antivirals are eligible if no evidence of active infection.
15. Class III or IV heart failure (as defined by the New York Heart Association - NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease within 6 months prior to Screening.
16. Cardiac arrhythmia not controlled by medical management.
17. Clinically significant thrombotic events within 6 months prior to leukapheresis and/or inability to stop anti-coagulation for at least 2 weeks prior to TAC01-HER2 infusion.
18. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, non-metastatic squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
19. Pregnant or lactating.
20. As determined by the Investigator, any uncontrolled medical, psychological, familial, sociological, or geographical condition(s) that do(es) not permit compliance with the protocol.
21. Participation in or has participated in a study using an investigational device within 4 weeks prior to study treatment..
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

    Combination Arm Only Specific Exclusions:
24. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
25. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-related AE (irAE).
26. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
27. Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of trial treatment.
28. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
29. Has history of an allogeneic stem cell transplant or a solid organ transplant.
30. Has a history of radiation pneumonitis. (Note: Cannot receive prior radiotherapy within 2 weeks of start of pembrolizumab. Note: Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation [≤2 weeks of radiotherapy] to non-CNS disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Lurie Cancer Center - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, Newark, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Sidney Kimmel Cancer Center - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal/Montreal Hospital University Center (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In addition to the 23 subjects who were assigned to groups, 5 additional subjects were enrolled but not not assigned to groups:
  * 3 died before group assignment
  * 2 failed to meet pre-treatment inclusion criteria
Groups:
- TAC01-HER2 DL1: Lymphodepletion followed by TAC01-HER2 as a single IV infusion, with a potential for a second dose administration.
  TAC01-HER2: 1-3x10^5 TAC01-HER2 and:
  * fludarabine and cyclophosphamide, or
  * cyclophosphamide
- TAC01-HER2 DL2: Lymphodepletion followed by TAC01-HER2 as a single IV infusion, with a potential for a second dose administration.
  TAC01-HER2: 6-8x10^5 TAC01-HER2 and:
  * fludarabine and cyclophosphamide, or
  * cyclophosphamide
- TAC01-HER2 DL3: Lymphodepletion followed by TAC01-HER2 as a single IV infusion, with a potential for a second dose administration.
  TAC01-HER2: 1-3x10^6 TAC01-HER2 and:
  * fludarabine and cyclophosphamide, or
  * cyclophosphamide
- TAC01-HER2 DL4: Lymphodepletion followed by TAC01-HER2 as a single IV infusion, with a potential for a second dose administration.
  TAC01-HER2: 6-8x10^6 TAC01-HER2 and:
  * fludarabine and cyclophosphamide, or
  * cyclophosphamide
- Unassigned: Not Treated
Period: Overall Study
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4 | Unassigned
Started | 4 | 4 | 3 | 12 | 5
Completed | 4 | 4 | 3 | 12 | 0
Not Completed | 0 | 0 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 3
Not completed — failed to meet pre-treatment inclusion criteria | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4 | Total
Number analyzed (Participants) | 4 | 4 | 3 | 12 | 23
Age, Continuous [Median (Full Range); unit: years] | 65.5 [50 to 68] | 61.5 [42 to 70] | 52 [40 to 63] | 59 [45 to 74] | 59 [40 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 9 | 15
  Male | 0 | 3 | 2 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 2 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 1 | 0 | 0 | 1
  Race: Black | 0 | 0 | 0 | 0 | 0
  Race: White | 4 | 3 | 3 | 11 | 21
  Race: Other | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — * 0: Fully active, able to carry on all pre-disease performance without restriction
  * 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 1 | 2 | 2 | 5 | 10
    1 | 3 | 2 | 1 | 7 | 13
Cancer type [Count of Participants; unit: Participants]
  Breast | 0 | 0 | 2 | 1 | 3
  Gastric | 1 | 1 | 0 | 4 | 6
  Other | 3 | 3 | 1 | 7 | 14
Stage of disease at screening [Count of Participants; unit: Participants] — * Stage III: The cancer has grown significantly and may have spread to distant lymph nodes.
  * Stage IV: The cancer has metastasized, meaning it has spread to other parts of the body.
  Participants
    Stage III | 0 | 0 | 0 | 1 | 1
    Stage IV | 4 | 3 | 2 | 10 | 19
    Unknown | 0 | 1 | 1 | 1 | 3
Bridging therapy [Count of Participants; unit: Participants] — Received bridging chemotherapy between enrollment and treatment
  Participants
    Yes | 2 | 1 | 0 | 10 | 13
    No | 2 | 3 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Incidence of Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as:
  * Grade 4 or 5 events determined by the Investigator to be related to the investigational product, with the exception of Grade 4 laboratory abnormalities that are rapidly reversible or correctable without substantial safety concerns.
  * Grade ≥3 TAC T cell-associated acute infusion reactions persisting for ≥24 hours
  * Grade ≥3 TAC T cell-associated CRS or neurotoxicity persisting for ≥72 hours
  * Grade ≥3 cardiovascular or pulmonary toxicity persisting for ≥72 hours
  * Grade ≥3 immune-related toxicities
  * Grade ≥3 organ toxicities or non-hematologic toxicities that do not improve to baseline within 7 days
  * Clinically consequential Grade ≥3 neutropenia or thrombocytopenia lasting ≥30 days from TAC01-HER2 administration. Clinically consequential is defined as febrile neutropenia, serious infection, or bleeding events.
Time Frame: 28 days
Population: One participant at DL4 was classified as non-evaluable due to a fatal aspiration pneumonia event (unrelated to TAC01-HER2) before the DLT period elapsed.
Measure: Count of Participants; unit: Participants
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 11
Participants
  Yes | 0 | 0 | 0 | 1
  No | 4 | 4 | 3 | 10

2. Secondary Outcome: Phase 1: Determine Recommended Phase 2 Dose (RP2D) for TAC01-HER2 Monotherapy
Description: RP2D was determined by the Data and Safety Monitoring Committee using the keyboard design method (<95% chance that the DLT rate exceeds 30%).
Time Frame: Up to 28 Days Post TAC01-HER2 infusion
Population: One subjects was classified as non-evaluable due to a fatal aspiration pneumonia event (unrelated to TAC01-HER2) before the period lapsed
Measure: Number; unit: TAC01-HER2 cells/kg
Groups:
- All Participants Who Received at Least One Dose of TAC01-HER2: All participants who received at least one dose of TAC01-HER2 (at DL1, DL2, DL3 and DL4)
Arm/Group | All Participants Who Received at Least One Dose of TAC01-HER2
Number analyzed (Participants) | 22
TAC01-HER2 cells/kg | 7000000

3. Secondary Outcome: Phase 1: Evaluate Overall Response Rate (ORR)
Description: Defined as the percentage of treated subjects with a complete or partial response (CR or PR) as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Time Frame: 24 months
Population: One subject at DL4 was classified as non-evaluable due to a fatal aspiration pneumonia event (unrelated to TAC01-HER2) before the first scheduled follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 11
Participants | 0 | 1 | 0 | 1

4. Secondary Outcome: Phase 1: Evaluate Duration of Response (DoR)
Description: Defined as time from first response to disease progression, end of study, start of another anticancer therapy, or death
Time Frame: 24 months
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 11
months | 0 [0 to 0] | 2.2 [2.2 to 2.2] | 0 [0 to 0] | 1.9 [1.9 to 1.9]

5. Secondary Outcome: Phase 1: Evaluate Overall Survival (OS)
Description: Defined as participants alive after 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 12
Participants | 2 | 4 | 1 | 7

6. Secondary Outcome: Phase 1: Evaluate Disease Control Rate (DCR)
Description: Defined as the percentage of treated subjects with stable disease (SD), PR, and CR as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST)Version 1.1.
Time Frame: 24 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 11
Participants | 0 | 3 | 2 | 6

7. Secondary Outcome: Phase 1: Progression-Free Survival (PFS) or Time to Progression (TTP)
Description: Defined as time from infusion to disease progression or death from any cause
Time Frame: 24 months
Population: One participant at DL2 withdrew consent before disease progression and was thus unevaluable for PFS.
Measure: Median (Full Range); unit: months
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 3 | 3 | 12
months | 0.9 [0.8 to 1] | 2.8 [0.9 to 12.4] | 2.6 [1 to 4.7] | 0.95 [0.1 to 3.2]

8. Secondary Outcome: Phase 1: Cmax of TAC01-HER2 (Pharmacokinetics; PK)
Description: Defined as the maximum concentration of TAC T cells after infusion; assessed by vector copy number
Time Frame: Pre-treatment, days 3, 4 or 5, 8, 11, 14 or15, 18, 21 or 22, 25, 29, 42, months 3, 6, 9, 12, 18, 24 or end of study, and at the confirmatory progressive disease visit
Population: One subject at DL4 was non-evaluable.
Measure: Median (Full Range); unit: vector copy number/μg gDNA
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 11
vector copy number/μg gDNA | 75.5 [39 to 853] | 247 [29 to 1640] | 63 [52 to 206] | 797 [202 to 5288]

9. Secondary Outcome: Phase 1 and Phase 2: Tmax of TAC01-HER2 (PK)
Description: Defined as the the first study day the Cmax is reached
Time Frame: as for outcome 8
Population: One subject at DL4 was non-evaluable.
Measure: Median (Full Range); unit: days after infusion
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4
Number analyzed (Participants) | 4 | 4 | 3 | 11
days after infusion | 4 [4 to 29] | 18.5 [11 to 22] | 15 [15 to 22] | 8 [8 to 22]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for a period of 90 days. All-Cause Mortality was assessed through study completion for each participant (for up to 2 years).
Arm/Group | TAC01-HER2 DL1 | TAC01-HER2 DL2 | TAC01-HER2 DL3 | TAC01-HER2 DL4 | Unassigned
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/4 | 2/3 | 5/12 | 4/5
Serious Adverse Events (participants affected / at risk) | 4/4 | 2/4 | 2/3 | 9/12 | 3/5
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/3 | 12/12 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAC01-HER2 DL1 (N=4) | TAC01-HER2 DL2 (N=4) | TAC01-HER2 DL3 (N=3) | TAC01-HER2 DL4 (N=12) | Unassigned (N=5)
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 2 | 0 | 1 | 1 | 3
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Partial Duodenal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Thromboembolic Event (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Transaminitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAC01-HER2 DL1 (N=4) | TAC01-HER2 DL2 (N=4) | TAC01-HER2 DL3 (N=3) | TAC01-HER2 DL4 (N=12) | Unassigned (N=5)
Leukopenia (Blood and lymphatic system disorders) | 4 | 4 | 0 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 1 | 8 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 5 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 3 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 4 | 0
Disease progression (General disorders) | 2 | 0 | 1 | 1 | 3
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Procedural pain (General disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 7 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Refeeding syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 3 | 11 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 4 | 0
Serum ferritin increased (Investigations) | 0 | 2 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood fibrinogen increased (Investigations) | 0 | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 3 | 1 | 3 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 3 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 5 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gallbladder oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Partial Duodenal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Thromboembolic Event (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Transaminitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs have the right to publish or discuss the results of the Study provided such disclosure is submitted to the SPONSOR for review and comment 45 days prior to submission for publication or 60 days prior to presentation. The PIs have agreed to defer disclosure at the request of the SPONSOR, to permit the filing of any desired patent applications. Any disclosure based on the results obtained at PI's Site shall not be made before the first multi-centre publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT04727151/Prot_SAP_000.pdf